CLINICAL TRIAL: NCT01172145
Title: Treatment of Apathy in Alzheimer's Disease With Modafinil
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Cephalon (Industry)
Responsible Party: Laura L. Frakey, Brown University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1F32MH075583-01 (NIH); 1F32MH075583-01 (NIH)
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Results first posted 2011-03-04 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2010-09

CONDITIONS: Apathy; Alzheimer's Disease
Keywords: apathy; Alzheimer's disease; activities of daily living performance; caregiver burden
MeSH Terms: conditions — Lethargy; Alzheimer Disease; Caregiver Burden | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cholinesterase inhibitor only (Placebo Comparator)
  Interventions: Drug: Placebo
- Cholinesterase Plus Modafinil (Experimental)
  Interventions: Drug: Modafinil

INTERVENTIONS:
Drug: Modafinil — 100 mg in the morning for the first week and 200 mg in the morning for the remaining seven weeks
  Other Names: Provigil
  Arms: Cholinesterase Plus Modafinil
Drug: Placebo — 100 mg in the morning for the first week and 200 mg in the morning for the remaining seven weeks
  Arms: Cholinesterase inhibitor only

SUMMARY:
This study examined the effects of modafinil on apathetic symptomatology, performance of activities of daily living (ADLs) and caregiver burden in individuals with Alzheimer's disease (AD).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mild to moderate stage Probable Alzheimer's disease
* on a stable dose of a cholinesterase inhibitor medication for at least 30 days
* clinically elevated levels of apathy as measured by the Frontal Systems Behavior Scale

Exclusion Criteria:

* diagnosis of Major Depression
* focal brain lesion on neuroimaging
* history of significant substance abuse
* history of significant head trauma with loss if consciousness >10 minutes

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-07; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura L Frakey, Ph.D., Principal Investigator — Memorial Hospital of Rhode Island
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Frakey LL, Salloway S, Buelow M, Malloy P. A randomized, double-blind, placebo-controlled trial of modafinil for the treatment of apathy in individuals with mild-to-moderate Alzheimer's disease. J Clin Psychiatry. 2012 Jun;73(6):796-801. doi: 10.4088/JCP.10m06708. Epub 2012 May 15. PMID 22687392

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a Memory Disorders Clinic and the community between 2005 and 2007
Groups:
- Cholinesterase Inhibitor Only: participants who received placebo
- Cholinesterase Plus Modafinil: participants who received modafinil (200 mg per day)
Period: Overall Study
Arm/Group | Cholinesterase Inhibitor Only | Cholinesterase Plus Modafinil
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cholinesterase Inhibitor Only | Cholinesterase Plus Modafinil | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 11 | 10 | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 79.36 (7.62) | 75.27 (8.34) | 77.32 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Apathy
Description: The Frontal Systems Behavior Scale. Raw scores are converted to T-Scores using published norms. T-Scores have a mean of 50 and a standard deviation of 10. T-scores less than or equal to 64 are within average range. T-scores equal to or greater than 65 are indicative of a clinically significant problem. Higher scores indicate greater problem severity.
Time Frame: at baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Cholinesterase Inhibitor Only | Cholinesterase Plus Modafinil
Number analyzed (Participants) | 11 | 11
T-score | 88.91 (11.95) | 95.64 (10.79)
Statistical Analysis 1: Comparison: Cholinesterase Inhibitor Only vs Cholinesterase Plus Modafinil; Test type: Superiority or Other; p = 0.181, t-test, 2 sided; Mean Difference (Final Values) = -1.385, 95% CI 2-sided [-16.86 to 3.40], Standard Error of Mean 4.86

2. Primary Outcome: Apathy
Description: The Frontal Systems Behavior Scale.Raw scores are converted to T-Scores using published norms. T-Scores have a mean of 50 and a standard deviation of 10. T-scores less than or equal to 64 are within the average range. T-scores equal to or greater than 65 are indicative of a clinically significant problem. Higher scores indicate greater problem severity.
Time Frame: after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Cholinesterase Inhibitor Only | Cholinesterase Plus Modafinil
Number analyzed (Participants) | 11 | 11
T-score | 82.09 (13.52) | 89.09 (9.61)

3. Secondary Outcome: Lawton Brody Activities of Daily Living Questionnaire
Description: Caregiver reported performance of personal and instrumental activities of daily living (ADLs. There are 6 personal ADLs (i.e. dressing, grooming, eating, etc) and 8 instrumental ADLs (i.e. managing finances, transportation, food preparation) which are assessed. Each item is awarded 2 points for fully independent, 1 point for minimal or moderate support required, and 0 points for full support. Maximum score for independence with all personal and instrumental ADL's is 28.
Time Frame: at baseline
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Cholinesterase Inhibitor Only | Cholinesterase Plus Modafinil
Number analyzed (Participants) | 11 | 11
raw score | 19.00 (5.25) | 16.18 (4.81)

4. Secondary Outcome: The Direct Assessment of Functional Status Scale
Description: A direct, examiner observed assessment of basic and instrumental activities of daily living. Participants are awarded points for correct performance of activities. Raw score is used for statistical comparison.
Time Frame: at baseline
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Cholinesterase Inhibitor Only | Cholinesterase Plus Modafinil
Number analyzed (Participants) | 11 | 11
raw score | 89.09 (7.84) | 84.55 (16.11)

5. Secondary Outcome: Zarit Burden Inventory
Description: Measure of Caregiver Burden. Caregiver rates each item assessing burden on a 0 to 4 point scale with higher numbers reflecting more frequent occurence of the behavior or feeling being assessed.
Time Frame: at baseline
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Cholinesterase Inhibitor Only | Cholinesterase Plus Modafinil
Number analyzed (Participants) | 11 | 11
raw score | 28.36 (21.09) | 31.18 (8.73)

6. Secondary Outcome: Lawton Brody Activities of Daily Living Questionnaire
Description: as for outcome 3
Time Frame: after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Cholinesterase Inhibitor Only | Cholinesterase Plus Modafinil
Number analyzed (Participants) | 11 | 11
raw score | 19.00 (5.54) | 15.64 (5.43)

7. Secondary Outcome: The Direct Assessment of Functional Status Scale
Description: as for outcome 4
Time Frame: after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Cholinesterase Inhibitor Only | Cholinesterase Plus Modafinil
Number analyzed (Participants) | 11 | 11
raw score | 88.36 (8.35) | 85.27 (14.16)

8. Secondary Outcome: Zarit Burden Inventory
Description: as for outcome 5
Time Frame: after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Cholinesterase Inhibitor Only | Cholinesterase Plus Modafinil
Number analyzed (Participants) | 11 | 11
raw score | 30.00 (20.56) | 30.00 (4.17)

ADVERSE EVENTS:
Arm/Group | Cholinesterase Inhibitor Only | Cholinesterase Plus Modafinil
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cholinesterase Inhibitor Only (N=11) | Cholinesterase Plus Modafinil (N=11)
Motor Tics (Nervous system disorders) | 0 (0) | 1 (1) — assessed by study neurologist

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No